CLINICAL TRIAL: NCT02825238
Title: The Effect of Hip and Core Muscle Strengthening on Pain, Function, Quality of Life and Movement Patterns in Persons With Patellofemoral Osteoarthritis: A Feasibility Study
Brief Title: Effect of Hip and Core Muscle Strengthening for Patellofemoral Osteoarthritis: A Feasibility Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of the Sciences in Philadelphia (Other)
Collaborators: University of Pennsylvania (Other); Thomas Jefferson University (Other)
Responsible Party: Principal Investigator, Lisa Hoglund, Associate Professor, University of the Sciences in Philadelphia
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 297090
Record Dates: First submitted 2016-06-29; First posted 2016-07-07 (Estimated); Last update posted 2018-05-08 (Actual); Status verified 2018-05

CONDITIONS: Patellofemoral Osteoarthritis
Keywords: exercise; osteoarthritis; knee; patellofemoral pain
MeSH Terms: conditions — Motor Activity; Osteoarthritis; Patellofemoral Pain Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention): Control group, did not undergo intervention.
- Exercise group (Experimental): Experimental, exercise group, underwent intervention
  Interventions: Other: Supervised exercise program

INTERVENTIONS:
Other: Supervised exercise program
  Arms: Exercise group

SUMMARY:
The purpose of this research is to develop and test the feasibility of an exercise intervention for persons with painful knee osteoarthritis involving the patella (kneecap). Participants in the patellofemoral osteoarthritis (PFOA) group will be treated with a 6-week supervised exercise program that targets strengthening the hip and trunk core muscles. Painfree control participants will attend one session to gather biomechanical, strength, and function data for use in comparison to the patellofemoral osteoarthritis group. Feasibility outcomes include adherence to the treatment program, recruitment, and retention. It is hypothesized that PFOA group participants will change score on a knee pain and function questionnaire by the minimum clinically important difference score for positive improvement at the end of the 6-week intervention program.

DETAILED DESCRIPTION:
The investigators propose to develop and test the feasibility of a 6-week supervised hip and core muscle exercise intervention for persons with painful patellofemoral osteoarthritis (PFOA), a common condition for middle-aged and older adults. Currently there is limited evidence regarding effective conservative interventions for PFOA, a chronic condition that is painful and limits function and quality of life. Exercise is recommended as a first-line treatment for knee osteoarthritis, but the optimal type of exercise for PFOA is unknown. This intervention is based upon similar programs shown to improve pain and function in younger persons with patellofemoral pain, a condition that may lead to PFOA. Feasibility outcomes include adherence to the treatment program, recruitment, retention, and the impact of the intervention on participants' pain and function at 6-weeks and 6 months after finishing the program. The investigators will also compare PFOA participants to a matched pain-free volunteer control group to explore the differences in their biomechanics, muscle strength, pain report, and function at baseline. Data from this feasibility study will be used to design a future randomized controlled trial investigating the efficacy of conservative exercise interventions for PFOA. The investigators' overarching goal is to develop a conservative exercise intervention that improves the symptoms, function, and quality of life of persons with PFOA.

ELIGIBILITY:
Inclusion Criteria:

Patellofemoral Osteoarthritis group: 1) age 35-70 years, 2) have been diagnosed with knee osteoarthritis in one or both knees with symptoms primarily in the anterior knee, 3) radiographic evidence of ≥ Grade 1 osteophytes or joint space narrowing at the patellofemoral joint according to the Osteoarthritis Research Society International (OARSI) grading scale (0 = none, 1 = mild/possible, 2 = moderate/definite, 3 = severe), 4) pain produced by ≥ 2 of the following: descending steps, ascending steps, sit-to-stand, squatting, kneeling, prolonged knee flexion, increased activity (e.g., hiking), morning stiffness < 30 minutes, stiffness after sitting ≥ 30 minutes, history of patellar subluxation or dislocation in the past.

Control group: 1) age 35-70 years, 2) no known diagnosis by a physician of knee osteoarthritis, 3) pain free in the lower extremities at the time of enrollment into the study and for 1 week prior to enrollment.

Exclusion Criteria:

Patellofemoral Osteoarthritis (PFOA) group: 1) the presence of other conditions that may cause knee pain (e.g., patellar tendonitis, rheumatoid arthritis), 2) neurologic or musculoskeletal conditions that may alter lower extremity kinematics (e.g., multiple sclerosis, hip arthritis/arthroplasty), 3) history of a fracture of the knee, 4) pregnancy, 5) knee injections within the past 3 months, 6) inability to understand English.

Control group: 1) all previously listed exclusion criteria for the PFOA group, 2) knee pain produced by 2 or more of the following: descending steps, ascending steps, sit-to-stand, squatting, kneeling, prolonged knee flexion, or a history of patellar subluxation or dislocation in the past.

Ages: 35 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2012-10-23 (Actual); Primary Completion 2015-12-11 (Actual); Study Completion 2015-12-11 (Actual)

PRIMARY OUTCOMES:
Feasibility (adherence) | 6 weeks
  Adherence to supervised program (≥ 80% complete 10 supervised exercise sessions and 2 data collection sessions): Percentage adherence.
Feasibility (retention rates) | 6 weeks
  Completion of baseline and 6-week evaluation sessions. Percentage completion for both data collection sessions.
Feasibility (follow-up response): questionnaire | 6 months
  Response to 6-month follow-up - return Knee Injury and Osteoarthritis Outcome Score (KOOS) questionnaire (≥ 80% complete and return KOOS): Percentage completion and return for KOOS.
Feasibility (recruitment rates) | 4 years
  Total number enrolled and total number screened out.
Feasibility (establish viability of underlying treatment model): global rating of change | 6 weeks
  Response to participation in intervention program in terms of overall rating of change (≥ 80% will achieve Global Rating of Change score ≥ 3 [scale -5 to 5] - positive numbers indicate positive change).
Feasibility (follow-up response): exercise diary | 6 months
  Response to 6-month follow-up - return exercise diary (≥ 80% complete and return exercise diary): Percentage completion and return for diary.
Feasibility (establish viability of underlying treatment model): pain rating | 6 weeks
  Response to participation in intervention program in terms of pain rating (≥ 80% will change score on KOOS pain subscale by the minimum clinically important difference score for positive improvement [positive change of 10 points] - at the end of the 6-week intervention program).
Feasibility (establish viability of underlying treatment model): activity of daily living rating | 6 weeks
  Response to participation in intervention program in terms of activity of daily living rating (≥ 80% will change score on KOOS activity of daily living (ADL) subscale by the minimum clinically important difference score for positive improvement [positive change of 10 points] - at the end of the 6-week intervention program).

SECONDARY OUTCOMES:
Establish impact of intervention on physical performance | 6 weeks
  Change in score on Timed-Up-and-Go test.
Determine long-term benefits of intervention: pain rating | 6 months
  Change in score of KOOS pain subscale score for positive improvement: 6-month follow-up KOOS versus baseline KOOS scores (more positive scores equals lower pain level)
Determine long-term benefits of intervention: activity of daily living rating | 6 months
  Change in score of KOOS ADL subscale score for positive improvement: 6-month follow-up KOOS versus baseline KOOS scores (more positive scores equals better function in activities of daily living)

OTHER OUTCOMES:
Change in peak isometric muscle torque: hip abductors, hip extensors, hip external rotators, and knee extensors | 6 weeks
Change in hip and knee joint biomechanics during step-down and sit-to-stand tasks | 6 weeks
Change in KOOS symptoms subscale | 6 weeks
Change in KOOS sport/recreation subscale | 6 weeks
Change in KOOS quality of life subscale | 6 weeks
Examine differences between patellofemoral osteoarthritis group and painfree control group in terms of lower extremity biomechanics (joint angles) | 6 weeks
  Lower extremity peak joint angles will be measured with a motion capture system during functional activities.
Examine differences between patellofemoral osteoarthritis group and painfree control group in terms of lower extremity muscle torque | 6 weeks
  Lower extremity peak isometric torque will be measured with a dynamometer (force gauge).
Examine differences between patellofemoral osteoarthritis group and painfree control group in terms of physical performance on the Timed-Up-and Go test | 6 weeks
  Time to perform the Timed-Up-and-Go test of walking ability will be measured with a stop watch.
Examine differences between patellofemoral osteoarthritis group and painfree control group in terms of symptoms on the Knee Injury and Osteoarthritis Score (KOOS) questionnaire | 6 weeks
  Responses to the KOOS questionnaire will be gathered and the score calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Lisa T Hoglund, PhD, PT, Principal Investigator — Thomas Jefferson University
Locations (2):
- United States (2):
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University of the Sciences, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Hoglund LT, Pontiggia L, Kelly JD 4th. A 6-week hip muscle strengthening and lumbopelvic-hip core stabilization program to improve pain, function, and quality of life in persons with patellofemoral osteoarthritis: a feasibility pilot study. Pilot Feasibility Stud. 2018 Apr 6;4:70. doi: 10.1186/s40814-018-0262-z. eCollection 2018. PMID 29636983
- See also: A 6-week hip muscle strengthening and lumbopelvic-hip core stabilization program to improve pain, function, and quality of life in persons with patellofemoral osteoarthritis: a feasibility pilot study. — https://pilotfeasibilitystudies.biomedcentral.com/articles/10.1186/s40814-018-0262-z